CLINICAL TRIAL: NCT04769830
Title: Study on the Value of Digital Continuous Bowel Sound Monitoring in AGI of Critically Ill Patients With ICU
Brief Title: Biomarkers and Bowel Sounds in Patients With Acute Gastrointestinal Injury
Acronym: BABSIPWAGI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2021LSK-013
Record Dates: First submitted 2021-02-06; First posted 2021-02-25 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-05

CONDITIONS: Gastrointestinal Injury
Keywords: biomarkers; Continuous bowel sound detection; Critically ill patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Citrulline，Intestinal fatty acid binding protein and so on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AGI group: Collect the characteristic data of intestinal sound, such as 24-hour average intestinal rate, duration of gastrointestinal sound, amplitude, maximum frequency, average frequency, etc., and detect citrulline, intestinal fatty acid binding protein and so on.
  Interventions: Other: Bowel sound
- non-AGI group: Collect the characteristic data of intestinal sound, such as 24-hour average intestinal rate, duration of gastrointestinal sound, amplitude, maximum frequency, average frequency, etc., and detect citrulline, intestinal fatty acid binding protein and so on.
  Interventions: Other: Bowel sound

INTERVENTIONS:
Other: Bowel sound — The characteristic data of bowel sounds, such as 24-hour average intestinal rate, duration of gastrointestinal sounds, amplitude, maximum frequency and average frequency, were collected to observe the differences of intestinal sounds among different AGI grades.

SUMMARY:
The incidence of gastrointestinal diseases is high in intensive care unit (intensive care unit,ICU). In critically ill patients, the intestinal tract is the "engine" of multiple organ dysfunction syndrome (Multiple organ dysfunction syndrome,MODS) and a component of multiple organ dysfunction syndrome, which is closely related to the poor prognosis of critically ill patients. In 2012, the abdominal working group of the European Association of critical Care Medicine (the European Society of Intensive Care Medicine,ESICM) put forward the concept of "acute gastrointestinal injury" (acute gastrointestinal injury,AGI), which was defined as gastrointestinal dysfunction caused by acute disease in critically ill patients. However, the grading system is complex and general, which does not reflect other gastrointestinal functions such as endocrine, immunity, barrier and so on, and lacks the support of objective laboratory results. When patients with acute gastrointestinal injury, gastrointestinal digestion and absorption, endocrine, immunity, barrier function are affected in varying degrees. The levels of indexes reflecting gastrointestinal digestion and absorption, endocrine and immunity were different among different AGI grades. The purpose of this study was to observe the characteristics of AGI bowel sounds in critically ill patients with ICU by digital continuous bowel sound monitoring, and to explore the clinical value of bowel sounds characteristics in AGI of critically ill patients combined with the changes of biomarkers of gastrointestinal injury.

DETAILED DESCRIPTION:
In this study, digital bowel sound monitoring equipment was used to continuously monitor the bowel sound of critically ill patients with ICU. This technology added the intestinal sound characteristic database to the data processing center, analyzed and identified the intestinal sound data through the intestinal sound recognition algorithm, further analyzed the parameters such as audio frequency, spectrum and power spectrum, and observed the changes of biomarkers such as citrulline and intestinal fatty acid binding protein.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old and ≤ 80 years old.
* The time of staying in ICU is expected to be more than 48 hours.
* The patient or legal guardian or legal representative signs the informed consent form.

Exclusion Criteria:

* It is estimated that the hospitalization time of ICU is less than 24 hours, and the case data are incomplete.
* Age > 80 years old; patients with chronic or primary gastrointestinal diseases (such as Crohn's disease, ulcerative colitis, gastrointestinal ulcer), short bowel syndrome, gastrointestinal surgery (history of partial or total gastrectomy), malignant tumor.
* Pregnant or lactating women.
* Patients with severe cardiovascular disease and hemodynamic instability may have cardiorespiratory arrest in a short period of time.
* The patient himself or the agent refused to sign the informed consent form or participate in another clinical trial.
* The researchers determined that other conditions in which the patient was not suitable for selection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The critically ill patients treated in the Department of intensive Care of the first affiliated Hospital of Xi'an Jiaotong University were selected as the sample source.
Sampling Method: Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-09-25 (Estimated); Study Completion 2022-09-25 (Estimated)

PRIMARY OUTCOMES:
Changes of 24-hour average intestinal sound rate | Days 1, 2, 3, 7
  Times per minute

SECONDARY OUTCOMES:
Changes of citrulline level | Days 1, 2, 3, 7
  μmol/L
Changes of intestinal fatty acid binding protein level | Days 1, 2, 3, 7
  ng/L
Changes of motilin level | Days 1, 2, 3, 7
  ng/L
Changes of gastrin level | Days 1, 2, 3, 7
  ng/L

CONTACTS AND LOCATIONS:
Overall Officials: Qindong Shi, Chief, Study Chair — Director of intensive Care Unit
Locations (1):
- First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi, China